CLINICAL TRIAL: NCT06424535
Title: Integrated Traditional Chinese and Western Medicine to Care for the Late Stage of Mild to Moderate Burns and Scalds
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CMUH113-REC1-055
Record Dates: First submitted 2024-05-07; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Burns and Scalds
Keywords: Acupuncture; Chinese medicine; Burns; Scalds; Low level laser
MeSH Terms: conditions — Burns | interventions — Medicine, Chinese Traditional

STUDY DESIGN:
Intervention Model Description: 1:1 randomized controlled crossover study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): 1. Traditional Chinese medicine for internal or external use
  2. Acupuncture or laser acupuncture treatment
  3. Acupoint massage
  4. Traditional Chinese Medicine Cake Acupoint Application:
  5. Nursing and health education and guidance
  6. Dietary hygiene education
  Interventions: Other: Chinese medicine for internal or external use、Acupuncture or Laser acupuncture pen treatment、Acupoint Tuina massage、Acupoint application of traditional Chinese herbal medicinal cake
- control group (Active Comparator): Routine Western medicine burn and scald care prescribed by department doctor
  Interventions: Other: Western medicine

INTERVENTIONS:
Other: Chinese medicine for internal or external use、Acupuncture or Laser acupuncture pen treatment、Acupoint Tuina massage、Acupoint application of traditional Chinese herbal medicinal cake — The treatment project a Chinese medicine practitioner based individual needs of the patient, and will be followed by a four-week treatment.
  1. Traditional Chinese medicine for internal or external use: prescribe Chinese medicine based on syndrome differentiation and treatment of the patient's condition.
  2. Acupuncture or laser acupuncture treatment: Traditional Chinese medicine practitioners select acupuncture points to treat based on the patient's condition, and treat them twice a week for 20 minutes each time.
  3. Acupoint massage: Select treatment acupoints and techniques according to the patient's condition, 20 minutes at a time.
  4. Traditional Chinese Medicine Cake Acupoint Application: Warm Navel Cream to the CV-4 (Guanyuan) acupoint once a day
  5. Nursing and health education and guidance
  6. Dietary hygiene education: personalized western nutrition and TCM dietary guidance suggestions based on TCM constitution syndromes.
  Other Names: Traditional Chinese medicine
  Arms: intervention group
Other: Western medicine — Patients will receive routine Western medicine treatments as per individual patient's needs. The medications and bandages can vary due to the depth and size of the burn and scald.
  Other Names: Routine Western medicine care
  Arms: control group

SUMMARY:
To explore the effectiveness of TCM interventional treatment in shortening the recovery time and improving accompanying symptoms of burns and scalds. A single-center, randomized control crossover trial will compare TCM intervention to routine western medicine intervention.

DETAILED DESCRIPTION:
Burns are an irreversible traumatic injury. When the skin suffers severe burns, it will cause a systemic shock to the individual. Although in recent years, with the advancement of medical technology, the mortality rate from burns and scalds has dropped significantly compared with the past, patients with burns and scalds also face many challenges during the treatment process, including having to endure the pain of the wound and the risk of infection during hospitalization. During the rehabilitation period after discharge, scarring, limb contracture, skin itching and appearance changes caused by burns and scalds will cause a significant decline in the patient's quality of life and lead to depression, withdrawal, social isolation and other phenomena. Traditional Chinese medicine is based on empirical medicine and the observation records of doctors. It has been passed down from generation to generation, and also have experience in treating fever. There are external and internal treatments for treating burns and scalds. External medicinal powders and ointments, such as Sanhuang powder,Jinchuang ointment,Ziyun ointment, etc. For internal medicine,Huanglian Jiedu Decoction,Qingying Decoction,Xijiao Dihuang Decoction,Tuoli Disinfection Powder,Shenling Baizhu Powder, etc. can be used according to different syndrome types. In addition, past studies have also confirmed that acupuncture can relieve burns and scalds and inhibit scar formation. Acupuncture can also improve gastrointestinal function and can be used to maintain good nutrient absorption in patients during the treatment of burns and scalds.

There are few large-scale studies on the joint treatment of burns and scalds between Chinese and Western medicine. Therefore, the purpose of this project is to compare the wound healing status and healing time between two groups that simply received conventional Western medicine treatment and conventional treatment plus interventional treatment with Chinese medicine. The study investigate traditional Chinese medicine interventional treatment model for mild to moderate burns and scalds, and hope to implement it clinically in the future to improve medical quality and treatment efficiency.

A single-center, randomized control crossover trial. This study will be conducted at the Burn and Scald Center and Plastic Surgery/Traditional Chinese Medicine Clinic of China Medical University Hospital. When patients seek medical treatment for burns and scalds, they will be evaluated by a plastic surgeon and randomly assigned into two groups. One group will receive conventional Western medicine treatment plus TCM intervention. Different treatment strategies will be adopted depending on the severity of the condition, and the first assessment will be conducted before TCM interventional treatment. , a post-test was conducted four weeks after treatment. Afterward, the two groups will be alternated. The group that did not receive TCM intervention received TCM interventional treatment for four weeks, while the other group received only conventional Western medicine treatment. The assessment items included: assessment of wound and pain status. Pain status was assessed using the Visual Analogue Scale (VAS), and scars were assessed using the Vancouver Scar Scale (VSS). Assess, and record critical indicators according to clinical needs, such as caloric requirement (kcal), daily fluid requirement (ml), daily urine output (ml) and other physiological parameters, and record the burn area (Modified Lund-Browder chart) and depth. The control group will be treated with conventional Western medicine. Outcome measurements will be assessed at baseline, 4 weeks, and 4 weeks after crossover (8 weeks). The goal of our study is to measure the effectiveness of TCM interventional treatment in shortening recovery time and improving accompanying symptoms of burns and scalds.

ELIGIBILITY:
Inclusion Criteria:

* Age：20-90.
* Patients with mild to moderate injuries and burns that meet the American Burn Association (ABA) injury classification.

Exclusion Criteria:

* Patients refuse TCM intervention.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | At baseline, 4 weeks, and 4 weeks after crossover (8 weeks)
  Measured by the Visual Analogue Scale (VAS) 0-10: 0 =No Pain 2 = Mild 4 = Nagging 6 =Miserable 8 =Intense 10 = Worst
Vancouver Scar Scale | At baseline, 4 weeks, and 4 weeks after crossover (8 weeks)
  Scars measurement will be assessed using the Vancouver Scar Scale (VSS)Each characteristic is given a score, which are added together to give an overall score between 0 and 13. Higher score indicate wrost outcome.

SECONDARY OUTCOMES:
Caloric intake per day | At baseline, 4 weeks, and 4 weeks after crossover (8 weeks)
  Amount of caloric (kcal) consumed per patient per day measured by department's nurse calculated by the amount of calories the patient consumed via feeding tube or oral feeding
Daily fluid requirement (ml) | At baseline, 4 weeks, and 4 weeks after crossover (8 weeks)
  Amount of daily fluid requirement (ml) per patient per day measured by department's nurse in milliliters (ml) of fluid intake and intravenous infusion or oral intake.
Daily urine output | At baseline, 4 weeks, and 4 weeks after crossover (8 weeks)
  Amount of Daily urine output measured by department's nurse in milliliters(ml) per patient patients Daily urine output measured by department's nurse in milliliters(ml) per day
Lund-Browder chart | At baseline, 4 weeks, and 4 weeks after crossover (8 weeks)
  burn area measured by Modified Lund-Browder chart, the score represents percentage (%) of the body cover by the burn along with body area, it score 0-100 and a higher score indicate worst outcome

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan